CLINICAL TRIAL: NCT03783286
Title: Nutritional Impact of Ivacaftor Treatment in 4 Month to 2 Year Old Children With CF Gating Mutations
Brief Title: Ivacaftor Treatment in 4 Month to 2 Year Old CF Subjects
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Principal Investigator, Virginia Stallings, Director of Nutrition Center Children's Hospital of Philadelphia, Professor of Pediatrics, Perelman School of Medicine at the University of Pennsylvania, Children's Hospital of Philadelphia
Other Study IDs: 18-015299
Record Dates: First submitted 2018-12-18; First posted 2018-12-21 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Cystic Fibrosis
Keywords: CF transmembrane conductance regulator; CFTR; Gating Mutations
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and stool collections
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ivacaftor — Ivacaftor (Kalydeco®, Vertex Pharmaceuticals Inc.) was the first of a new class of drugs that improved CFTR gating dysfunction (2, 3, 4). For such mutations (G551D, G178R, S549N, S549R, G551S, G970R, G1244E, S1251N, S1255P, G1349D) that permit CFTR expression at the cell membrane but compromise its activity.
  Other Names: Kalydeco

SUMMARY:
The purpose of this research study is to determine the effects of clinically prescribed ivacaftor treatment on 4-24 month old children with CF and gating mutations on sleeping energy expenditure, growth status and gut health and function.

DETAILED DESCRIPTION:
Ivacaftor is a novel FDA approved therapy for patients with CF and gating mutations who are 4 months and older. This investigator-Initiated study is designed to evaluate the nutritional, growth and GI impact of ivacaftor treatment for the youngest (4-24 months) patient cohort and for whom FDA approval has recently been granted. This proposal directly extends the previous highly informative nutrition and weight gain investigation of ivacaftor treatment in the older patient cohort (1). The primary aims of the study are to evaluate the impact of 12 weeks of ivacaftor treatment in 4-24 month old subjects with CF and gating mutations on sleeping energy expenditure, growth status and gut health and function in 18 children with protocol evaluations at baseline (pre-treatment) and 6 and 12 weeks after clinically prescribed ivacaftor treatment has begun. Other outcomes of significant clinical interest in young subjects with CF will be explored. All subjects will be evaluated at the Children's Hospital of Philadelphia (CHOP) and will be recruited both regionally and nationally to ensure timely enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis with at least one CFTR gating mutation (E56K, G178R, S549R, S977F, F1074L, 2789+5G→A,P67L, E193K, G551D, F1052V, D1152H, 3272-26A→G, R74W, L206W, G551S, K1060T, G1244E, 3849+10kbC→T, D110E, R347H, D579G, A1067T, S1251N, D110H, R352Q, 711+3A→G, G1069R, S1255P, R117C, A455E, E831X, R1070Q, D1270N, R117H, S549N, S945L, R1070W, G1349D) approved for treatment
* Age: 4-24 months of age
* In their usual state of good health
* A clinical decision has been made for subject to begin ivacaftor treatment
* Family committed to the 4 to 6 month study protocol with visits to CHOP that will last 2 or 3 days for the baseline visit (Visit 1) prior to ivacaftor and the 12 week visit (Visit 3) after clinically prescribed ivacaftor treatment has begun, and will last 2 days for the 6 week visit (Visit 2) after ivacaftor treatment has begun.

Exclusion Criteria:

* On parenteral nutrition
* Use of any medications which are as inhibitors or inducers of cytochrome P450 (CYP) 3A
* Liver function tests elevated above 3x the reference range for age and sex
* Other illness affecting growth or nutritional status
* Other contraindications described for ivacaftor therapy

Ages: 4 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 4-24 month old subjects with a diagnosis of cystic fibrosis with at least one CFTR gating mutation of these ten (G551D, G178R, S549N, S549R, G551S, G1244E, S1251N, S1255P, G1439D, or R117H) approved for treatment in a usual state of good health with a clinical decision to start ivacaftor treatment.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Sleeping Energy Expenditure | 12 Weeks
  Investigators will examine the effects of 12 weeks of Ivacaftor treatment on subject's SEE. Using indirect calorimetry, SEE will be assessed using a computerized metabolic cart Vmax ENCORE at each protocol visit while the child is asleep. SEE will be assessed in the morning if possible and careful note of previous feeding of the child, including the time of day, amount of food, and feeding interval prior to test
Anthropometric Assessment | 12 Weeks
  Investigators will examine the effects of 12 weeks of Ivacaftor treatment on subject's BMI. Investigators will compare the results to BMI Z scores over 12 weeks compared to baseline.

SECONDARY OUTCOMES:
Fecal Elastase I/Pancreatic Function | 12 Weeks
  Investigators will examine the effects of 12 weeks of Ivacaftor treatment on subject's pancreatic function. Pancreatic function will be assessed at two visits by obtaining spot stool samples with fecal elastase 1. The concentration of fecal elastase I is indicative of pancreatic function.
Fecal Calprotectin/Gut Inflammation | 12 Weeks
  Investigators will examine the effects of 12 weeks of Ivacaftor treatment on subject's gut health and function. Spot stool samples will be obtained to determine fecal calprotectin, a marker for gut inflammation.
Plasma Total Fatty Acids: | 4 to 6 months
  Investigators will examine the effects of 12 weeks of Ivacaftor treatment on subject's dietary fat absorption. A total plasma fatty acid panel will be assessed to measure the change in status of 22 fatty acids, the concentration of plasma fatty acids is indicative of dietary fat absorption.

OTHER OUTCOMES:
Dietary Intake | 12 Weeks
  Three day weighed food record will be obtained and to determine changes in dietary caloric intake and micro and macronutrient intake over the course of 12 weeks on ivacaftor treatment. The weighed food in grams will be used to determine the calories consumed, as well as calories from fat. The caloric intake will be used to determine micro and macro nutrient intake.
Serum fat soluble vitamins A, D, E and K, bile acids, and serum calprotectin | 12 Weeks
  Investigators will examine the changes in serum vitamin A, E, D and K concentrations after 12 weeks of Ivacaftor treatment. Additionally, investigators will examine the changes in total serum bile acids concentration and 14 bile acid species. Additionally, serum calprotectin will be obtained as a marker of lung and gut inflammation.
Muscle/Fat Stores | 12 Weeks
  Investigators will measure body composition to determine muscle and fat store changes over the course of 12 weeks on ivacaftor treatment compared to baseline.
Growth Status/Growth Velocity | 12 Weeks
  Investigators will observe the changes in growth status/growth velocity. This will be assessed amongst three different measurements- length (cm), weight (kg) and head circumference (cm). Each value will be used to calculate the growth velocity percentile of the subjects over the course of 12 weeks on ivacaftor treatment compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Stallings, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stallings VA, Sainath N, Oberle M, Bertolaso C, Schall JI. Energy Balance and Mechanisms of Weight Gain with Ivacaftor Treatment of Cystic Fibrosis Gating Mutations. J Pediatr. 2018 Oct;201:229-237.e4. doi: 10.1016/j.jpeds.2018.05.018. Epub 2018 Jul 18. PMID 30029855
- [Background] Van Goor F, Hadida S, Grootenhuis PD, Burton B, Cao D, Neuberger T, Turnbull A, Singh A, Joubran J, Hazlewood A, Zhou J, McCartney J, Arumugam V, Decker C, Yang J, Young C, Olson ER, Wine JJ, Frizzell RA, Ashlock M, Negulescu P. Rescue of CF airway epithelial cell function in vitro by a CFTR potentiator, VX-770. Proc Natl Acad Sci U S A. 2009 Nov 3;106(44):18825-30. doi: 10.1073/pnas.0904709106. Epub 2009 Oct 21. PMID 19846789
- [Background] Accurso FJ, Rowe SM, Clancy JP, Boyle MP, Dunitz JM, Durie PR, Sagel SD, Hornick DB, Konstan MW, Donaldson SH, Moss RB, Pilewski JM, Rubenstein RC, Uluer AZ, Aitken ML, Freedman SD, Rose LM, Mayer-Hamblett N, Dong Q, Zha J, Stone AJ, Olson ER, Ordonez CL, Campbell PW, Ashlock MA, Ramsey BW. Effect of VX-770 in persons with cystic fibrosis and the G551D-CFTR mutation. N Engl J Med. 2010 Nov 18;363(21):1991-2003. doi: 10.1056/NEJMoa0909825. PMID 21083385
- [Background] Ramsey BW, Davies J, McElvaney NG, Tullis E, Bell SC, Drevinek P, Griese M, McKone EF, Wainwright CE, Konstan MW, Moss R, Ratjen F, Sermet-Gaudelus I, Rowe SM, Dong Q, Rodriguez S, Yen K, Ordonez C, Elborn JS; VX08-770-102 Study Group. A CFTR potentiator in patients with cystic fibrosis and the G551D mutation. N Engl J Med. 2011 Nov 3;365(18):1663-72. doi: 10.1056/NEJMoa1105185. PMID 22047557
- [Background] Energy and protein requirements. Report of a joint FAO/WHO/UNU Expert Consultation. World Health Organ Tech Rep Ser. 1985;724:1-206. No abstract available. PMID 3937340
- [Background] Schofield WN. Predicting basal metabolic rate, new standards and review of previous work. Hum Nutr Clin Nutr. 1985;39 Suppl 1:5-41. PMID 4044297
- [Background] 7. World Health Organization. WHO Child Growth Standards: Length/height-for-age, weight-for-age, weight-for-length, weight-for-height, and body mass index-for-age. Geneva, Switzerland: WHO Press, World Health Organization; 2006.
- [Background] Borowitz D, Baker SS, Duffy L, Baker RD, Fitzpatrick L, Gyamfi J, Jarembek K. Use of fecal elastase-1 to classify pancreatic status in patients with cystic fibrosis. J Pediatr. 2004 Sep;145(3):322-6. doi: 10.1016/j.jpeds.2004.04.049. PMID 15343184
- [Background] Borowitz D, Lin R, Baker SS. Comparison of monoclonal and polyclonal ELISAs for fecal elastase in patients with cystic fibrosis and pancreatic insufficiency. J Pediatr Gastroenterol Nutr. 2007 Feb;44(2):219-23. doi: 10.1097/MPG.0b013e31802c41de. PMID 17255835
- [Background] O'Connor MG, Seegmiller A. The effects of ivacaftor on CF fatty acid metabolism: An analysis from the GOAL study. J Cyst Fibros. 2017 Jan;16(1):132-138. doi: 10.1016/j.jcf.2016.07.006. Epub 2016 Jul 26. PMID 27473897
- [Background] 11. World Health Organization. WHO Child Growth Standards: Head circumference-for-age, arm circumference-for-age, triceps skinfold-for-age, and subscapular skinfold-for-age. Geneva, Switzerland: WHO Press, World Health Organization; 2007.
- [Background] 12. WHO Multicenter Growth Reference Study Group. WHO Child Growth Standards: Growth Velocity Based on Weight, Length and Head Circumference: Methods and Development. Geneva, Switzerland: WHO Press: World Health Organization; 2009.
- [Derived] Tindall A, Bass R, Maqbool A, Stallings VA. Changes in nutrition and growth status in young children in the first 12 weeks of ivacaftor therapy. J Cyst Fibros. 2023 Nov;22(6):989-995. doi: 10.1016/j.jcf.2023.04.010. Epub 2023 Jul 10. PMID 37438197

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT03783286/Prot_SAP_003.pdf
  • Informed Consent Form (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT03783286/ICF_002.pdf